CLINICAL TRIAL: NCT02929212
Title: Effect of Number of Meals on Metabolism After Weight Loss Surgery
Acronym: LAF 28
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Blandine Laferrere, Professor of Medicine, Columbia University, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AAAO3051; R01DK067561 (NIH)
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Morbid Obesity
Keywords: Gastric Bypass; Meal Texture; Meal Number; GLP-1; Glucose
MeSH Terms: conditions — Obesity, Morbid | interventions — Acetaminophen; Single Person; Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Solid Meal Study Group A (Other): Patients Pre and Post-GBP who are randomly assigned to receive solid meals on study days given as one, 600 kcal, meal.
  Interventions: Other: Solid Meal; Drug: Acetaminophen; Other: Single, 600 kcal meal
- Liquid Meal Study Group A (Other): Patients Pre and Post-GBP who are randomly assigned to receive liquid meals on meal study days, given as one, 600 kcal, meal
  Interventions: Other: Liquid Meal; Drug: Acetaminophen; Other: Single, 600 kcal meal
- Solid Meal Study Group B (Other): Patients Pre and Post-GBP who are randomly assigned to receive solid meals on study days given as three, 200 kcal, meals.
  Interventions: Other: Solid Meal; Drug: Acetaminophen; Other: Multiple, 200 kcal meals
- Liquid Meal Study Group B (Other): Patients Pre and Post-GBP who are randomly assigned to receive liquid meals on meal study days, given as three, 200 kcal, meals.
  Interventions: Other: Liquid Meal; Drug: Acetaminophen; Other: Multiple, 200 kcal meals

INTERVENTIONS:
Other: Solid Meal — Subjects will receive solid meals during meal study
  Arms: Solid Meal Study Group A; Solid Meal Study Group B
Other: Liquid Meal — Subjects will receive liquid meals, during meal study
  Arms: Liquid Meal Study Group A; Liquid Meal Study Group B
Drug: Acetaminophen — All subjects given acetaminophen to measure gastric emptying
Other: Single, 600 kcal meal — Subjects will receive a single, 600 kcal meal during meal study
  Arms: Liquid Meal Study Group A; Solid Meal Study Group A
Other: Multiple, 200 kcal meals — Subjects will receive three, 200 kcal meals, during meal study
  Arms: Liquid Meal Study Group B; Solid Meal Study Group B

SUMMARY:
The purpose of this study is to determine the effect of meal size and texture on the levels of incretin hormone, GLP-1, after Gastric Bypass Surgery (GBP). Patterns of food intake change after bariatric surgery and patients often eat multiple small low-calorie meals, a pattern that may affect blood glucose as well as incretin levels. Whether the release of GLP-1 after an oral challenge or a single liquid meal has any physiological relevance in 'real life' setting of multiple small meals diet is unclear.

DETAILED DESCRIPTION:
The main goal is to study the effect of meal size and texture on incretin levels after GBP. Patients will be studied before GBP (T0) and 12-15 months after GBP (T1). At T0 and T1, patients will come for 2 study days for 8 hours: On one study day, a single meal will be served, on the second study day, three small meals, with the order of the conditions randomly assigned. The total amount of calories (600 kcal) and the over all nutrient composition (55% CHO, 15 % protein, 30% fat) will be equivalent between conditions. The meals will be either all solid or all liquid. Patients enrolled in the study will be randomly assigned to solid or liquid test meals.

Recruitment and data gathering for this study were performed at St. Luke's Hospital in New York, NY. Data Analysis was performed at Columbia University Medical Center in New York, NY.

ELIGIBILITY:
Inclusion Criteria: morbidly obese individuals, BMI above 35 and less than 50 kg/m2 who chose GBP as treatment for their obesity

* Must be able to attend all study visits at St. Luke's Roosevelt Hospital Center in Manhattan, New York City
* Individuals with or without Type 2 Diabetes Mellitus are eligible

Exclusion Criteria:

* Patients with abnormal thyroid, renal function, known malabsorption syndrome or a seizure disorder requiring anti epileptic therapy, and/or elevation of liver enzymes three times above the normal limit.
* Patients with intestinal conditions such as chronic diarrhea, diverticulitis, or irritable bowel syndrome.
* Currently pregnant or nursing.
* Known cardiovascular disease.
* Patient with current mucosal (gastrointestinal, respiratory, urogenital) or skin (cellulitis) infection
* Any other condition which, in the opinion of the investigators, may make the candidate unsuitable for participation in this study.
* past history of severe food allergy
* History of Type 1 Diabetes Mellitus
* Individuals taking insulin, thiazolidinedione, exenatide, or DPP-IV inhibitors

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Difference in GLP-1 levels before and after gastric bypass surgery | 12-15 months
  Investigators will assess GLP-1 levels in subjects pre and post-GBP
Difference in glucose levels before and after gastric bypass surgery | 12-15 months
  Investigators will assess glucose in subjects pre and post-GBP
Difference in insulin levels before and after gastric bypass surgery | 12-15 months
  Investigators will assess insulin levels in subjects pre and post-GBP

SECONDARY OUTCOMES:
Difference in GLP-1 levels in solid vs liquid meals | 12-15 months
  Investigators will assess GLP-1 levels in subjects eating either liquid or solid meals at both pre-surgery and post-surgery time points
Difference in glucose levels in solid vs liquid meals | 12-15 months
  Investigators will assess glucose levels in subjects eating either liquid or solid meals at both pre-surgery and post-surgery time points
Difference in insulin levels in solid vs liquid meals | 12-15 months
  Investigators will assess insulin levels in subjects eating either liquid or solid meals at both pre-surgery and post-surgery time points

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, Principal Investigator — Columbia University
Locations (1):
- New York Obesity Nutrition Research Center, St. Luke's-Roosevelt Hospital Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No